CLINICAL TRIAL: NCT01045226
Title: A Phase II Trial of Proton Radiation Therapy of Using Standard Fractionation for Low-and Low-Intermediate Risk Adenocarcinoma of the Prostate
Brief Title: Proton Radiation Therapy in Treating Patients With Prostate Cancer
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: participants are no longer being followed up.
Sponsor: Abramson Cancer Center at Penn Medicine (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: UPCC 08809; NCI-2009-01500
Record Dates: First submitted 2010-01-05; First posted 2010-01-08 (Estimated); Last update posted 2023-02-01 (Actual); Status verified 2023-01

CONDITIONS: Prostate Cancer
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Proton Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Arm I (Experimental): Patients undergo proton radiotherapy once daily 5 days a week for approximately 9 weeks in the absence of disease progression or unacceptable toxicity.
  Interventions: Procedure: Proton Beam Radiation Therapy; Other: Quality-of-Life assessment; Other: Questionnaire Administration

INTERVENTIONS:
Procedure: Proton Beam Radiation Therapy — Proton Beam Radiation Therapy
Other: Quality-of-Life assessment — Quality of Life Assessment
Other: Questionnaire Administration — Questionnaire Administration

SUMMARY:
RATIONALE: Specialized radiation therapy that delivers a high dose of radiation directly to the tumor may kill more tumor cells and cause less damage to normal tissue.

PURPOSE: This clinical trial is studying how well proton radiation therapy works in treating patients with prostate cancer.

DETAILED DESCRIPTION:
Detailed Description

PRIMARY OBJECTIVES:

I. Feasibility of proton radiation therapy (RT) using standard fractionation.

SECONDARY OBJECTIVES:

I. To determine freedom from failure (FFF) (vs. biochemical/clinical progression-free survival) with standard fractionation.

II. To determine the incidence of grade 2 or greater GU and GI toxicity with this regimen at 6 months, 2 years and 3 years.

III. To assess quality of life issues following completion of radiation therapy at 6 months and at 2 years.

IV. To assess incidence of impotence after the use of proton therapy at 3 years.

V. To determine freedom from biochemical failure (BF) at 5 years.

VI. To determine clinical failure: local and/or distant at 5 years. VII. To determine salvage androgen deprivation (SAD) use at 5 years. VIII. To determine progression free survival: using clinical, biochemical and SAD as events at 5 years.

IX. To determine overall survival at 5 years. X. To determine disease-specific survival at 5 years.

XI. Estimate prostate and normal structures movement during RT with the use of scans.

XII. Correlate pathologic and radiologic findings with outcomes at 5 years. XIII. Correlate PSA and free PSA levels with outcomes at 5 years. XIV. Correlate testosterone levels and variation with proton therapy and outcomes at 5 years.

XV. Develop a quality assurance process for proton prostate therapy.

OUTLINE:

Patients undergo proton radiotherapy once daily 5 days a week for approximately 9 weeks in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed at 3 months, every 6 months for 5 years, and then annually thereafter.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed prostate adenocarcinoma within 365 days of registration
* Clinical stages T1a-T2a N0 M0
* For any pelvic lymph node >= 1.5cm, biopsy of the lymph node is mandatory
* Histological evaluation of prostate biopsy with assignment of a Gleason score to the biopsy material; Gleason score must be in the range 2-6; > 6 cores is strongly recommended; the highest Gleason score in any core reported on the pathology report will be used for determining inclusion
* PSA values < 10 ng/ml within 90 days prior to registration, done either prior to prostate biopsy or at least 21 days after prostate biopsy.
* Alkaline phosphatase within 60 days prior to registration. If alkaline phosphatase is elevated > 2 x the upper limit of institutional normal (UNL), patient must have radiological correlation to assess for metastases
* Zubrod status 0-1 documented within 60 days of registration
* Prior androgen deprivation is allowed; however, androgen deprivation will not be continued concurrently or as an adjuvant therapy
* Patients must give IRB-approved study-specific informed consent
* Patients must complete all required tests listed within the specified time frames
* Patients must be able to start treatment within 56 days of registration
* Members of all races and ethnic groups are eligible for this trial

Exclusion Criteria:

* Clinical stages T2c or greater
* PSA of 10 ng/ml or greater
* Gleason score 7 or higher
* Evidence of distant metastasis
* Evidence of lymph node involvement
* Previous prostate cancer surgery to include: prostatectomy, hyperthermia and cryosurgery
* Previous pelvic radiation for prostate cancer
* Androgen deprivation therapy prior to radiation is allowed; however, it is not acceptable if continued during radiation or as adjuvant therapy
* Active rectal diverticulitis, Crohn's disease, or ulcerative colitis are not allowed
* Prior systemic chemotherapy for prostate cancer
* History of proximal urethral stricture requiring dilatation

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Actual)
Dates: Start 2009-08 (Actual); Primary Completion 2020-12 (Actual); Study Completion 2022-03-17 (Actual)

PRIMARY OUTCOMES:
As a feasibility precaution patients will be treated and followed for a minimum of 60 days after completion of radiotherapy to determine feasibility | 5 years
Acute toxicity as assessed by NCI CTC Version 3.0 | 90 days

SECONDARY OUTCOMES:
Late toxicity as assessed by RTOG/EORTC late morbidity scoring system | 90 days
Biochemical/clinical progression-free survival | Time from start of radiotherapy to either documented increase in PSA or clinical progression of disease, death due to any cause or last patient contact alive

CONTACTS AND LOCATIONS:
Locations (1):
- Abramson Cancer Center of the University of Pennsylvania, Philadelphia, Pennsylvania, United States